CLINICAL TRIAL: NCT04108650
Title: Portuguese Version of the Fit & Strong! Program for Older Adults With Osteoarthritis
Brief Title: Portuguese Fit & Strong! for Older Adults With Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Instituto de Ciências Biomédicas Abel Salazar (ICBAS) (Unknown); Centro de Investigação em Tecnologias e Serviços de Saúde (Other); Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: F&S/111533/2015
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2020-11

CONDITIONS: Osteoarthritis
Keywords: Physical Activity; Health Education; Fit & Strong!
MeSH Terms: conditions — Osteoarthritis; Motor Activity; Health Education

STUDY DESIGN:
Who Masked: Participant
Masking Description: Experimental and control group had no interaction to each other during the study. For data collection was used an individual interview in a place that guarantee privacy. None participant were aware about the group that they will be allocated before the baseline assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fit & Strong! group (Experimental): The experimental group (23 participants) was enrolled in the intervention, the Fit & Strong! program. The program consists in 24 sessions each divided in two parts. The first part is the exercise component (60 minutes) and the second is the educational component (30 minutes). The program was provided in two classes, the first class took place from October to December 2017 and the second class took place from October to November 2018. The experimental group was enrolled in the intervention (8 weeks).
  Interventions: Other: Fit & Strong! group
- Control group (No Intervention): To participants in the control group (8 participants) were offered the possibility of enrolling in the program the following year after posttest measurement for both the intervention and control groups was complete.

INTERVENTIONS:
Other: Fit & Strong! group — Consistent with the original format of F&S!, the classes met three times per week for 90 minutes each for 8 weeks (24 sessions in total). Each class session consisted of 60 minutes of exercise and 30 minutes of health education. The exercise protocol included 10 minutes of warm-up and cool-down exercises, 20 minutes of low-intensity aerobic exercises, and 20 minutes of lower extremity strengthening exercises. The health education program focused on symptom management and behavioral strategies to increase physical activity and commitment to lifestyle change.
  Arms: Fit & Strong! group

SUMMARY:
Fit & Strong! (F&S!) is a non-pharmacological intervention designed for older people with osteoarthritis with proven efficacy. This program was developed and implemented among American patients. It is composed by two components: physical exercise with health education. In total, the program last eight weeks, and meets three times per week (24 sessions), for 90 minutes per session. The nationals and internationals statistics showed that Portugal has a high prevalence of OA, in particular in the knee or hip. Considering this fact and the negative impact in OA patients' lives the F&S! program was culturally adapted for Portugal, which constitutes its first formal adaptation to an international population and setting.

Therefore, a randomized controlled trial was developed to the effects of F&S! among Portuguese older adults with lower-extremity OA, particularly, with respect to physical performance (walking speed, balance, lower body strength), pain, stiffness, functionality, physical activity, anxiety, depression and fear of movement. Participants were identified and referred from the electronic medical record maintained by general practitioners in Health Care Centers. Participants were randomly allocated to the experimental or to the control and were assessed three times (baseline, posttest and 4-months follow-up). Data analysis included descriptive statistics (medians and interquartile ranges) to describe participants' characteristics. The comparison between the experimental and the control group at baseline was performed using the Mann-Whitney U test for continuous variables and the Fisher test for categorical variables. Within each group, changes over time (pretest, posttest, follow-up) were analyzed using the Wilcoxon signed-rank test. Between group comparisons of differences in outcome variables between pretest, posttest and 4-month follow-up were analyzed using the Mann-Whitney U test.

DETAILED DESCRIPTION:
Fit & Strong! (F&S!) is an evidence-based intervention for OA in the U.S. developed at the University of Illinois, Chicago. This program was designed for older adults who have lower extremity joint pain and stiffness caused by OA. It is a pioneer multi-component intervention that incorporates physical exercise with health education for long lasting behavior change. The intervention last 8 weeks, and meets three times per week (24 sessions), for 90 minutes per session. Each session includes one hour of stretching, low-impact aerobics/ fitness walking, and strengthening exercises using adjustable ankle cuff weights and exercise bands, and balance exercises. The class was structured to begin with a warm-up activity, then, an aerobic activity and balance exercises, strengthening exercises, end a cold down activity with stretching and relaxation exercises were performed. The last 30 minutes of each session include structured, manual-based group discussion/health education. The educational component aims to facilitate symptom management, increase confidence in ability to exercise, and commitment to lifestyle change. Toward the end of the eight weeks, each participant meets individually with the instructor to develop a tailored adherence contract (a core element of the program). Participants received a "Participant Manual" with the description of the all program and the logs that have to fill during the program.

In Portugal, similar to other developed countries, the prevalence of OA is high. It is estimated that the self-reported prevalence of knee OA in adults 18 years and older was 11.1%, 5.9% in men and 14.2% in women. Rates of hip OA were 5.5%, 2.2% in men and 7.4% in women. The National Rheumatic Diseases Observatory (ONDOR) that based its findings on radiographic evidence, found a prevalence of knee OA in adults 40 years of age or older of 56.9% in men and 57.7% in women; radiographic hip OA was 54.8% in men and 24.5% in women.

Considering the high prevalence and the negative impact that OA has on patients' lives, in contrast to the positive effects demonstrated by F&S! in U.S., the program was culturally adapted in Portugal, which constitutes its first formal adaptation to an international population and setting. Therefore, a randomized controlled trial was developed to analyze the effects of the Portuguese version of the F&S!. This study sought to analyze the effects of F&S! among Portuguese older adults with lower-extremity OA, particularly, with respect to physical performance (walking speed, balance, lower body strength), pain, stiffness, functionality, physical activity, anxiety, depression and fear of movement.

Participants were identified and referred from the electronic medical record maintained by general practitioners in Health Care Centers.This phase of the study was conducted in two waves: the first wave lasted for three months (May 2017 to July 2017) and the second took place over five months (March 2018 to July 2018). After the identification of the potential participants by general practitioners, the principal investigator contacted the potential participants by phone to reinforce the invitation and to schedule a face-to-face interview (baseline assessment). During the phone contact an eligibility screen was used to confirm the presence of inclusion/exclusion criteria. Participants were randomly allocated by the researcher to the experimental or to the control group after the baseline assessment.

We used face-to-face interviews to collect the data in three distinct moments: baseline, posttest (at the end of the program) and 4-months follow up. Experimental group was enrolled in the Portuguese F&S! Program. The program was provided in two classes, the first class took place from October to December 2017 and the second class took place from October to November 2018.

Thirty one participants who were eligible and consented to participate, using a 2:1 randomization scheme, 23 participants were assigned to the experimental group and eight to the control group.

Regarding the data analysis, the descriptive statistics, including medians and the interquartile ranges were used to describe participant characteristics. The comparison between the experimental and the control group at baseline was performed using the Mann-Whitney U test for continuous variables and the Fisher test for categorical variables.

Within each group, changes over time (pretest, posttest, follow-up) were analyzed using the Wilcoxon signed-rank test. Between group comparisons of differences in outcome variables between pretest, posttest and 4-month follow-up were analyzed using the Mann-Whitney U test. Participants with an attendance rate of less than 50% were included in the baseline analyses but then were considered to be drop-outs and were excluded from posterior analyses. Results from these analyses are presented as medians and IQRs. Statistical analyses were performed using the Statistical Package for the Social Sciences for Windows (SPSS, version 25, IBM) and α=0.05 was used to determine significance level.

ELIGIBILITY:
Inclusion Criteria:

* age 50 years or older,
* lower extremity OA diagnosed according to the clinical criteria of the American College of Rheumatology (ACR) [14,15], and
* doctor's authorization to participate.

Exclusion Criteria:

* no recent (<6 months) joint replacements,
* no steroid injections in the last 3 months,
* no moderate to severe cognitive impairment,
* no rheumatoid arthritis,
* no diabetes mellitus and/or uncontrolled hypertension,
* no other health condition for which multicomponent physical exercise is not recommended.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Change in Physical Performance measured at baseline and posttest | 2 months
  The Short Physical Performance Battery was used to assess the physical performance. The Short Physical Performance Battery comprises a set of objective measures of lower extremity physical performance, including walking speed, chair-stands test, and balance test. Each physical performance measure was categorized into scale from 0 to 4, with 0 representing inability to do the test and 4 representing the highest level of performance. The scores of the three measures were summed with a score ranging from 0 to 12 and a higher score indicating better performance.
Change in Physical Performance measured at baseline and 4-months follow-up | 4 months
  The Short Physical Performance Battery was used to assess the physical performance. The Short Physical Performance Battery comprises a set of objective measures of lower extremity physical performance, including walking speed, chair-stands test, and balance test. Each physical performance measure was categorized into scale from 0 to 4, with 0 representing inability to do the test and 4 representing the highest level of performance. The scores of the three measures were summed with a score ranging from 0 to 12 and a higher score indicating better performance.
Change in pain measured at baseline and posttest | 2 months
  Pain was assessed by the Knee Injury and Osteoarthritis Outcome Score for people with knee OA; and by Hip disability and Osteoarthritis Outcome for people with hip OA. A score for each dimension is calculated as the sum of the items that are included, which is then converted to a 0-100 scale in which 0 represents extreme problems and 100 represents no problems.
Change in pain measured at baseline and 4-months follow-up | 4 months
  Pain was assessed by the Knee Injury and Osteoarthritis Outcome Score for people with knee OA; and by Hip disability and Osteoarthritis Outcome for people with hip OA. A score for each dimension is calculated as the sum of the items that are included, which is then converted to a 0-100 scale in which 0 represents extreme problems and 100 represents no problems.
Change in stiffness measured at baseline and posttest | 2 months
  Stiffness was assessed by the Knee Injury and Osteoarthritis Outcome Score for people with knee OA; and by Hip disability and Osteoarthritis Outcome for people with hip OA. A score for each dimension is calculated as the sum of the items that are included, which is then converted to a 0-100 scale in which 0 represents extreme problems and 100 represents no problems.
Change in stiffness measured at baseline and 4-months follow-up | 4 months
  Stiffness was assessed by the Knee Injury and Osteoarthritis Outcome Score for people with knee OA; and by Hip disability and Osteoarthritis Outcome for people with hip OA. A score for each dimension is calculated as the sum of the items that are included, which is then converted to a 0-100 scale in which 0 represents extreme problems and 100 represents no problems.
Change in functionality measured at baseline and posttest | 2 months
  Functionality was assessed by the Knee Injury and Osteoarthritis Outcome Score for people with knee OA; and by Hip disability and Osteoarthritis Outcome for people with hip OA. A score for each dimension is calculated as the sum of the items that are included, which is then converted to a 0-100 scale in which 0 represents extreme problems and 100 represents no problems.
Change in functionality measured at baseline and 4-months follow-up | 4 months
  Functionality was assessed by the Knee Injury and Osteoarthritis Outcome Score for people with knee OA; and by Hip disability and Osteoarthritis Outcome for people with hip OA. A score for each dimension is calculated as the sum of the items that are included, which is then converted to a 0-100 scale in which 0 represents extreme problems and 100 represents no problems.
Change in moderate and vigorous physical activity measured at baseline and posttest | 2 months
  Physical activity was assessed by International Physical Activity Questionnaire. This instrument provides information on time spent walking, in vigorous and moderate intensity activity and in sedentary activity. The scale consists of six questions: the number of days on which vigorous physical activity was performed in the previous seven days and the usual duration of such activity; the number of days on which moderate physical activity was performed in the previous seven days and the usual duration of such activity; and the number of days on which the person walked for at least 10 minutes in the previous seven days and the usual duration of walking.
Change in moderate and vigorous physical activity measured at baseline and 4-month follow-up | 4 months
  Physical activity was assessed by International Physical Activity Questionnaire. This instrument provides information on time spent walking, in vigorous and moderate intensity activity and in sedentary activity. The scale consists of six questions: the number of days on which vigorous physical activity was performed in the previous seven days and the usual duration of such activity; the number of days on which moderate physical activity was performed in the previous seven days and the usual duration of such activity; and the number of days on which the person walked for at least 10 minutes in the previous seven days and the usual duration of walking.
Change in depression and anxiety symptoms measured baseline and posttest | 2 months
  Depression and anxiety were assessed by the Hospital Anxiety and Depression Scale. It includes 14 items, seven of which assess anxiety and seven of which assess depression. Each item is scored on a four-point scale (from 0 to 3), with possible scores for each subscale (anxiety and depression) ranging from 0 to 21 points. A score of 11 or higher indicates the probable presence of the mood disorder.
Change in depression and anxiety symptoms measured baseline and 4-months follow-up | 4 months
  Depression and anxiety were assessed by the Hospital Anxiety and Depression Scale. It includes 14 items, seven of which assess anxiety and seven of which assess depression. Each item is scored on a four-point scale (from 0 to 3), with possible scores for each subscale (anxiety and depression) ranging from 0 to 21 points. A score of 11 or higher indicates the probable presence of the mood disorder.
Change in fear of movement measured at baseline and posttest | 2 months
  Fear of movement was assessed by the Brief Fear of Movement Scale. This instrument consists of 6 items scored on a 4-point scale from "strongly agree" to "strongly disagree". Higher scores indicate higher fear of movement.
Change in fear of movement measured at baseline and 4-months follow-up | 4 months
  Fear of movement was assessed by the Brief Fear of Movement Scale. This instrument consists of 6 items scored on a 4-point scale from "strongly agree" to "strongly disagree". Higher scores indicate higher fear of movement.

OTHER OUTCOMES:
Age | Baseline (Day 0)
  A structured interview was used to collect data, including age (continuous).
Sex | Baseline (Day 0)
  A structured interview was used to collect data, including sex (woman/man).
Marital Status | Baseline (Day 0)
  A structured interview was used to collect data, including marital status (with partner - married or living with; or without partner - windowed or divorced).
Labor participation | Baseline (Day 0)
  A structured interview was used to collect data, including current labor participation (employed, retired or unemployed).

CONTACTS AND LOCATIONS:
Overall Officials: Natália Duarte, Master, Principal Investigator — ICBAS, CINTESIS, University of Porto
Locations (1):
- Instituto de Ciências Biomédicas Abel Salazar, Universidade do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duarte N, Hughes SL, Paul C. Cultural adaptation and specifics of the Fit & Strong! program in Portugal. Transl Behav Med. 2019 Jan 1;9(1):67-75. doi: 10.1093/tbm/iby003. PMID 29546428
- [Background] Hughes SL, Seymour RB, Campbell R, Pollak N, Huber G, Sharma L. Impact of the fit and strong intervention on older adults with osteoarthritis. Gerontologist. 2004 Apr;44(2):217-28. doi: 10.1093/geront/44.2.217. PMID 15075418
- [Background] Hughes SL, Seymour RB, Campbell RT, Desai P, Huber G, Chang HJ. Fit and Strong!: bolstering maintenance of physical activity among older adults with lower-extremity osteoarthritis. Am J Health Behav. 2010 Nov-Dec;34(6):750-63. doi: 10.5993/ajhb.34.6.10. PMID 20604699
- [Background] Hughes SL, Seymour RB, Campbell RT, Huber G, Pollak N, Sharma L, Desai P. Long-term impact of Fit and Strong! on older adults with osteoarthritis. Gerontologist. 2006 Dec;46(6):801-14. doi: 10.1093/geront/46.6.801. PMID 17169935